CLINICAL TRIAL: NCT01692054
Title: Prediction and Detection of Intermediate and Long-term Developmental Hazards in Adolescents After Alcohol Intoxication
Brief Title: Risk and Protective Factors of Children and Adolescents Who Were Hospitalized Due to Alcohol Intoxication
Acronym: RiScA
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: IIA5-2511DSM220
Record Dates: First submitted 2012-08-21; First posted 2012-09-25 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Alcohol Use Disorders
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Alcohol intoxicated adolescents: Adolescents who were hospitalized due to acute alcohol intoxication
- Control group: adolescents who were hospitalized due to other medical conditions but not alcohol intoxication

SUMMARY:
The aim of the study is to improve the prognosis of the development of alcohol consumption by considering a variety of biological, psychological and social risk and protective factors. Therefore, young people who have been hospitalized due to acute alcohol intoxication within the past 5 to 12 years will be interviewed in order to assess aspects of healthy or impaired psychosocial development. The study will also include a control group of young adults who were in hospital due to other medical conditions. The identification of relevant cases will be based on medical records of several children's hospitals. These records will be analysed with regard to potential predictors of developmental hazards and protective factors.

ELIGIBILITY:
experimental group:

Inclusion Criteria:

* male and female volunteers who were hospitalized due to acute alcohol intoxication from January 1, 2000 to December 31, 2006
* written informed consent by the subject
* minimum age of 20 years

Exclusion Criteria:

* incapability to conduct interview

control group:

Inclusion Criteria:

* male and female volunteers who were hospitalized due to other medical conditions but not acute alcohol intoxication from January 1, 2000 to December 31, 2006
* written informed consent by the subject
* minimum age of 20 years

Exclusion Criteria:

* incapability to conduct interview

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: young adults living in Germany who were hospitalized due to alcohol intoxication (experimental group) or other medical conditions (control group) 5 to 12 years ago
Sampling Method: Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Alcohol Use Disorders | 5 to 13 years
  Alcohol Use Disorders as measured by the The Alcohol Use Disorders Identification Test

SECONDARY OUTCOMES:
Self-efficacy | 5 to 13 years
Life Satisfaction | 5 to 13 years

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Zimmermann, Dr, Principal Investigator — Universitaetsklinikum Carl Gustav Carus at the Technische Universitaet Dresden
Locations (1):
- Universitaetsklinikum Carl Gustav Carus at the Technische Universitaet Dresden, Dresden, Saxony, Germany